CLINICAL TRIAL: NCT04048941
Title: One Needle Hand Acupuncture (Combined) With Movement for Treatment of Musculoskeletal Disorders: A Blinded Randomized Controlled Trial Involving 3 Groups
Brief Title: One Needle Hand Acupuncture for MSK Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201904173
Record Dates: First submitted 2019-07-10; First posted 2019-08-07 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Acupuncture; Pain; Range of Motion
MeSH Terms: conditions — Pain | interventions — Movement

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Verum Acupuncture with Movement (Experimental): Verum acupuncture along radial side of 2nd metacarpal, following by active movement of previously painful body part x 10 minutes.
  Interventions: Procedure: One Needle Hand Acupuncture with Movement
- Verum Acupuncture without Movement (Active Comparator): Verum acupuncture along radial side of 2nd metacarpal, following by laying on examination table x 10 minutes.
  Interventions: Procedure: One Needle Hand Acupuncture without Movement
- Control Acupuncture with Movement (Sham Comparator): Sham/control acupuncture at acupoint LI4, following by active movement of previously painful body part x 10 minutes.
  Interventions: Procedure: Control Acupuncture with Movement

INTERVENTIONS:
Procedure: One Needle Hand Acupuncture with Movement — One needle is inserted along the radial aspect of the 2nd metacarpal which relieves pain at a distant site. Then, the subject is asked to perform a series of movements that were previously painful.
  Arms: Verum Acupuncture with Movement
Procedure: One Needle Hand Acupuncture without Movement — One needle is inserted along the radial aspect of the 2nd metacarpal which relieves pain at a distant site. Then, the subject is asked to lay quietly on the examination table.
  Arms: Verum Acupuncture without Movement
Procedure: Control Acupuncture with Movement — Control acupuncture at acupoint LI4 is performed, which should not have a large affect on pain at a distant site. Then, the subject is asked to perform a series of movements that were previously painful.
  Arms: Control Acupuncture with Movement

SUMMARY:
The purpose of this research study is to study the method of acupuncture called one needle hand acupuncture, where a needle is placed just in your hand, in order to treat pain in various locations. Benefits of acupuncture will be studied over time to determine short and long term effects of acupuncture, and see how acupuncture may alter or modify a patient's disease process.

DETAILED DESCRIPTION:
Patients with neck, shoulder, low back, or hip pain that is exacerbated by movement will be randomized 1:1:1 to receive either verum hand acupuncture at the correct location (with or without movement) or control acupuncture at a nearby incorrect location. After needling and as part of the intervention, the movement groups will perform gentle active range of motion (ROM) exercises, while the without movement group will lay on the examination table, all for 10 minutes. Immediately pre- and post- intervention, numeric pain rating scores (NPRS) and goniometer- or inclinometer-obtained ROM measurements will be recorded for the most provocative movement plane.

In the physical therapy literature, within-session improvements in pain and ROM have been shown to correlate with between-session improvements.All patients will complete PROMIS Pain Interference, Physical Function, Anxiety, and Depression measures prior to the acupuncture intervention and then 1,2, 4, and 8 weeks later.

Four potential treatment response modifiers will be assessed. In Traditional Chinese Medicine (TCM), a strong needling sensation felt by the patient during an acupuncture treatment is called a "deqi" response and is thought to be a positive prognostic sign. In Western medicine, a local twitch response (LTR) observed during needling of muscle trigger points is thought to represent a polysynaptic reflex and has been linked to local pain improvements.Other potential modifiers include patients' underlying musculoskeletal structural diagnosis and the provider's experience performing acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* Primary pain localized to neck, shoulder, low back, hip.
* Pain >=4 on Numeric Pain Rating Scale with one of predetermined motions.
* Willing to participate in study and fill out questionnaires.

Exclusion Criteria:

* Fracture, malignancy
* Condition that requires urgent treatment (e.g. cervical myelopathy)
* Contraindications to needling (e.g. pregnancy, active infection)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Numeric Pain Rating Scale (NPRS) | Pre-acupuncture, post-acupuncture + 10 minutes
  Change in Numeric Pain Rating Scale from Baseline. Range is -10 to +6 by increments of 1. NPRS of later time point minus NPRS at baseline with lower number being better.
Percentage Change in Pain | Immediately post-acupuncture, post-acupuncture + 10 minutes
  Percentage Change in Pain after Needling Treatment. Options are 0%, 25%, 50%, 75%, 100%. Patient reported outcome at 2 time points with higher percentage indicating more improvement and being better.

SECONDARY OUTCOMES:
Change in Total Arc of Motion | Pre-Acupuncture, post-acupuncture + 10 minutes
  Total Arc of Motion is defined as Painful Range of Motion + Reciprocal Range of Motion. Cervical motion include active flexion + extension, active left rotation + right rotation, active left sidebend + right sidebend. Lumbar motions include active flexion + extension, active left rotation + right rotation, active left sidebend + right sidebend. Shoulder motions include active flexion + extension, active abduction + cross arm adduction, passive external rotation with arm down at the side + internal rotation behind the back, passive external rotation with the shoulder abducted to 90 + internal rotation with the shoulder abducted to 90. Hip motions include active flexion + extension with knee straight, passive flexion and extension with the knee bent to 90, passive internal rotation with the hip flexed to 90 + external rotation with the hip flexed to 90. Measurements in degrees with range from 0 to 360, the larger the change in total arc of motion the better.

OTHER OUTCOMES:
Change in Patient-Reported Outcome Measurement Information Systems (PROMIS) | Pre-Acupuncture, 1 week post-acupuncture, 2 weeks post-acupuncture, 4 weeks post-acupuncture, 8 weeks post-acupuncture
  PROMIS is a computerized adaptive testing that our institution administers that provides patient reported measures in the domains of pain interference, physical function, anxiety, and depression. PROMIS scores are normalized to the general population with a mean of 50 and a standard deviation of 10. Range is 0 - 100. A decrease in pain interference, increase in physical function, decrease in anxiety, and decrease in depression is good with larger absolute changes being better.
Presence of Deqi response | During Acupuncture treatment
  Yes or No whether patient reported an ache, numbness, fullness, or electric sensation with needling.
Presence of Local twitch response | During Acupuncture treatment
  Yes or No whether provider observed/felt twitch in the hand with acupuncture needling.
Structural diagnosis | Pre-acupuncture
  Patient's structural diagnosis given by provider.
Change in RAND 12 score | Pre-acupuncture, 4 weeks post-acupuncture
  The RAND 12 is a brief health survey comprised of 12 items that looks at general health, and is broken up into physical health summary and mental health summary; Scores are calculated via computer and compared with a large database of patients; average score for US population is 50 with a standard deviation of 10

CONTACTS AND LOCATIONS:
Overall Officials: Tonia Thompson, Study Director — Washington University School of Medicine
Locations (1):
- Washington University Orthopedic Center, Chesterfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No